CLINICAL TRIAL: NCT04271384
Title: Stereotactic Ablative Radiotherapy in Combination With Nivolumab for Early-Stage Operable Non-Small Cell Lung Cancer: a Phase 2 Study
Brief Title: Stereotactic Ablative Radiotherapy With Nivolumab for Early-Stage Operable Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NivoSABR
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer Stage I
Keywords: Non-small cell lung cancer; nivolumab; pd-1; radiotherapy; stereotactic body radiotherapy; radiosurgery; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SABR + Nivolumab (Experimental): Pre-operative treatment with standard SABR (3 x 18 Gy or 5 x 10 Gy or 8 x 7.5 Gy) concomitant with nivolumab at 360 mg every 21 days x3 doses.
  Standard-of-care surgery to be performed after 12 weeks from D1 of treatment.
  Interventions: Combination Product: nivolumab

INTERVENTIONS:
Combination Product: nivolumab — Combined neoadjuvant therapy consisting of nivolumab + SABR
  Other Names: stereotactic ablative radiotherapy

SUMMARY:
Stage 1 non-small cell lung cancer (NSCLC) carries up to 30% chance of relapse in 5 years. This a phase 2 study that aims to determine the pathological complete response of the combination of stereotactic ablative radiotherapy (SABR) plus nivolumab as neoadjuvant treatment in early-stage non-small cell lung cancer. The patients will receive standard SABR + nivolumab at a dose of 360 mg every 21 days for 3 doses. The patient will undergo surgery 10 weeks after the last radiotherapy dose.

DETAILED DESCRIPTION:
Stage 1 non-small cell lung cancer (NSCLC) carries up to 30% chance of relapse in 5 years. Surgery is standard-of-care for this population. For patients who are not candidate for surgery, stereotactic ablative radiotherapy (SABR) is standard, with good local control but locoregional and distant failure. The use of preoperative SABR leads to a pathological complete response rate (pCR) of 60%. Anti-PD-1 has the ability to provoke a pCR in around 20% of patients as a single agent. Moreover, it has synergic activity with radiotherapy.

This a phase 2 study that aims to determine the pathological complete response of the combination of stereotactic ablative radiotherapy plus nivolumab as neoadjuvant treatment in early-stage non-small cell lung cancer. The patients will receive standard SABR, given either as 3, 5 or 8 fractions (depending on tumor size and location) + nivolumab at a dose of 360 mg every 21 days for 3 doses. The patient will undergo surgery 10 weeks after the last radiotherapy dose. We will measure translational biomarkers associated with either pCR or resistance to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Non-small cell lung carcinoma (NSCLC), with longest diameter measuring up to 4 cm, restricted to one pulmonary lobe, with no clinical lymph node involvement through PET-CT and/or invasive staging, when indicated (not mandatory in patients with cT1-T2a and no uptake in lymph nodes through PET-CT);
2. No previous treatment;
3. Lesion susceptible to treatment with SABR, based on imaging evaluation by radiation oncologist;
4. Good clinical surgery conditions (lung function test with an appropriate forced expiratory volume in one second [FEV1] and predicted post-operative FEV1 of 30% or higher), and lesion resectability, based on evaluation by a thoracic surgery team;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1 - Appendix C: Criteria for Performance Status evaluation.
6. Aged ≥ 18 years old.
7. Absence of immunosuppressive diseases, or autoimmune diseases on active treatment or with systemic treatment within the last 2 years, or conditions requiring use of immunosuppressive agents, or on corticotherapy at dose > 10 mg of prednisone or equivalent;
8. Agreement with having all biomarkers of the study analyzed, including fresh biopsy tumor tissue, if needed.
9. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for following completion of therapy for 5 months if female and 7 months if male. Female subjects of child- bearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
10. Patients must have an appropriate organic function evaluation within 4 weeks before recruitment, evidenced by:

    * Hemoglobin ≥ 9.0 g/dL
    * Leucometry > 2,000/mm3
    * Absolute neutrophil count ≥ 1,000/mm3
    * Platelet count ≥ 100,000/mm3
    * Creatinine clearance ≥ 30 mL/min.
    * Total bilirubin < 3 x upper limit of normal (ULN), except for patients with known Gilbert's syndrome.
    * Aspartate aminotransferase (AST) < 3,0 x ULN.
    * Alanine aminotransferase (ALT) < 3,0 x ULN.

Exclusion Criteria:

1. Patients with contraindication to surgical treatment due to lack of medical conditions or deterioration of clinical state.
2. Patients with any known or suspected active autoimmune diseases. Patients with vitiligo, type 1 diabetes mellitus, controlled autoimmune hypothyroidism, psoriasis with no need of systemic treatment, or other controlled conditions may be recruited.
3. Patients with conditions requiring use of corticosteroids at doses > prednisone 10 mg/day (or equivalent) or use of other immunosuppressive medications within 28 days before anticipated start of study drug. Inhaled corticoids are permitted, if needed.
4. Patients with any known active chronic liver condition.
5. Patients with history of previous malignancy treatment with curative intention within the last 2 years, except for in situ skin basal cell carcinoma and squamous cell carcinoma, which will be allowed. Patients with other malignancies not meeting the previous criteria may be considered for recruitment if the disease in question does not represent a competitive cause for death or has a low potential of progressing to metastatic disease. Patients with these conditions may be recruited if approved after review by the principal investigator.
6. Patients with known positivity for human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS) or any test positive for hepatitis B or hepatitis C virus representing non-eradicated active acute or chronic disease.
7. Previous treatment with anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibodies, or any other specific antibody or drug targeting T-cell co-stimulation or immune checkpoint pathways.
8. Major surgery within 28 days before the first dose of the study drug.
9. Exposure to previous thoracic radiation therapy before the first dose of the study drug.
10. Prisoners or subjects who are involuntarily incarcerated.
11. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
12. Known pregnancy or refusal of appropriate contraception in females with child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Pathologic complete response (pCR) after Pre-operative therapy | 12 weeks after first day of neoadjuvant therapy
  pCR is defined as absence of viable tumor cells after neoadjuvant therapy, evaluated on surgical specimen

SECONDARY OUTCOMES:
Major pathological response (MPR) | 12 weeks after first day of neoadjuvant therapy
  MPR will be defined as <10% of viable tumor cells
Safety: Treatment-related adverse events with continuous toxicity measure as per CTCAE v4.0 | Every 21 days during the 3 doses of nivolumab and during a 100-day period after the last dose of study-treatment
  Treatment safety will be evaluated as per CTCAE v4.0
Objective response rate (ORR) | At 10 (+/- 2) weeks after treatment start.
  ORR will be evaluated as per RECIST v1.1
Relapse-free survival (RFS) at 12 months | 12-month rate
  Relapse-free survival will be measured from the enrollment date until the date of radiological progression, unequivocal clinical progression or death.
Overall survival (OS) | 12-month rate
  OS will be measured on the date of treatment D1 until date of death (regardless of cause)
Resectability Rate | From baseline to the day of surgery (12+-2 weeks)
  Rate of complete surgical resections after study treatment
30-day surgical mortality | 30 days after surgery
  Proportion of patients alive after 30 days from surgical resection
Number of pathologic positive lymph nodes | From baseline to the day of surgery (12+-2 weeks)
  Number of pathologic lymph nodes that were clinically negative and were found to be positive after surgery
Correlated translational endpoints | Baseline and at surgery
  The following will be evaluated: mutation profile, transcriptome, immunohistochemical profile, and inflammatory infiltrate by flow cytometry from peripheral blood. Flow cytometry will be repeated for all patients in the surgical specimen and peripheral blood. The mutation profile, transcriptome and immunohistochemical profile will be repeated for patients who do not reach a pathological complete response in viable cells to evaluate for potential resistance mechanisms. The intestinal microbiome will be sequenced before and after treatment and correlated with the endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Schvartsman, MD, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No